CLINICAL TRIAL: NCT02759861
Title: A Phase IV, Single Arm, Open-Label Study to Determine the Efficacy and Safety of Ledipasvir/Sofosbuvir (LDV/SOF) in Treatment-Naive Alcoholic Subjects With Chronic Genotype 1 Hepatitis C Infection
Brief Title: Determine the Efficacy and Safety of Harvoni in Genotype 1 Chronic Hepatitis c Infected People Who Are Alcoholics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0121-16-FB
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Results first posted 2023-02-23 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Genotype 1 Hepatitis C Virus
MeSH Terms: interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Harvoni x 8 or 12 weeks (Experimental): patient will receive 8 or 12 weeks depending on clinical data
  Interventions: Drug: harvoni

INTERVENTIONS:
Drug: harvoni — 8 or 12 weeks of harvoni therapy with monthly nursing visiting to monitor alcohol and adherence of harvoni therapy
  Other Names: Ledipasvir/Sofosbuvir

SUMMARY:
To determine the efficacy and safety of Harvoni in treatment-naïve alcoholic subjects with Genotype 1 HCV infection

DETAILED DESCRIPTION:
determine the cure rate of Harvoni in treatment naïve alcoholic subjects with Genotype 1 HCV infection

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be willingly and able to provide written informed consent
2. Age 19 years of age or older (The age of consent in Nebraska)
3. HCV treatment-naïve, as defined as no prior exposure to any Interferon (IFN), RBV, or other FDA approved or experimental HCV-specific direct-acting antiviral agent
4. HCV RNA level at most 6 months prior to the Baseline/Day 1 visit.
5. HCV genotyping 1a, 1b, or mixed 1a/ab. Any non-definitive results will exclude the subject from study participation.
6. Alcohol misuse as defined by the Alcohol Use Disorders Identification Test (AUDIT) score subjects must score > 8 (associated with harmful or hazardous drinking)
7. Cirrhosis determination [up to 20% of study subjects may have cirrhosis]:

   1. Cirrhosis is defined as any one of the following:

      * History of a liver biopsy showing cirrhosis (e.g. Metavir score = 4 or Ishak score > 5)
      * Fibroscan showing cirrhosis or results > 12.5 kPa
      * FIBRO Spect II index consistent with F3 or F4 AND an AST : platelet ration index (APRI) of > 2 during Screening
   2. Absence of cirrhosis is defined as any one of the following:

      * Liver biopsy within 2 years of Screening showing absence of cirrhosis
      * Fibroscan within 6 months of Baseline/Day1 with a result of ≤ 12.5 kPa
      * FIBRO Spect II Index consistent with F0- F2 AND APRI of ≤ 1 during Screening
8. Liver imaging within 6 months of Baseline/Day 1 to exclude hepatocellular carcinoma HCC) is required
9. Subjects must have the following laboratory parameters at screening:

   1. ALT < 10 x the upper limit of normal (ULN)
   2. AST < 10 x ULN
   3. Direct bilirubin < 2.0 x ULN
   4. Platelets > 50,000
   5. HbA1c < 8.5%
   6. Creatinine clearance (CLcr) ≥ 60 mL /min, as calculated by the Cockcroft-Gault equation
   7. Hemoglobin ≥ 11 g/dL for female subjects; ≥ 12 g/dL for male subjects.
   8. Albumin ≥ 2.5 g/dL
   9. INR ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR.
10. Subject has not been treated with any investigational drug or device within 30 days of the screening visit.

Exclusion Criteria:

1. Pregnant women and nursing mothers are ineligible due to the possible risk of adverse effects in the newborn. Eligible patients of reproductive potential should use adequate contraception if sexually active.
2. Serious concurrent medical illness which would jeopardize the ability of the subject to receive the therapy as outlined in this protocol with reasonable safety.
3. Malignancy diagnosed or treated within 5 years (recent localized treatment of squamous or non-invasive basal cell skin cancers is permitted; cervical carcinoma in situ is allowed if appropriately treated prior to screening); subjects under evaluation for a malignancy are not eligible.
4. Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
5. Use of any prohibited concomitant medications within 30 days of the Baseline/Day 1 visit.
6. Known hypersensitivity to LDV/SOF

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mailliard, MD, Principal Investigator — UNMC
Locations (1):
- University of Nebraska, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Harvoni x 8 or 12 Weeks: patient will receive 8 or 12 weeks depending on clinical data
  harvoni: 8 or 12 weeks of harvoni therapy with monthly nursing visit to monitor alcohol and adherence of harvoni therapy
Period: Overall Study
Arm/Group | Harvoni x 8 or 12 Weeks
Started | 16
Completed | 15
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Harvoni x 8 or 12 Weeks
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 14
  Black | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Who Achieve Negative RNA in Alcoholics
Description: Sustained viral response in treatment -naive heavy alcohol drinking patients.
Time Frame: 12 weeks after the end of Harvoni therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Harvoni x 8 or 12 Weeks
Number analyzed (Participants) | 15
Participants | 14

2. Secondary Outcome: Number of Subjects With Advanced Fibrosis Score of F3/F4 Who Achieve SVR
Description: Number of alcoholics with HCV type 1 genotype who had advanced fibrosis F3/F4 who achieve SVR
Time Frame: 12 weeks after the end of Harvoni therapy
Population: Had fibrosis F3/F4
Measure: Count of Participants; unit: Participants
Groups:
- F3/F4: Subjects who had advances fibrosis F3/F4 who achieved SVR at 12 weeks
Arm/Group | F3/F4
Number analyzed (Participants) | 9
Participants | 8

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: All-Cause Mortality was assessed in the total enrolled population while the Serious and Other (Not including Serious) adverse events were assessed in the completed population.
Arm/Group | Harvoni x 8 or 12 Weeks
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 13/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harvoni x 8 or 12 Weeks (N=15)
Fatigue (General disorders) | 7 (7)
Headache (General disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Agitation (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT02759861/Prot_SAP_000.pdf